CLINICAL TRIAL: NCT03400891
Title: A Randomised Controlled Trial of a Program Based on the Theory of Planned Behaviour to Promote Fruit and Vegetables Intake Among Children. PROFRUVE Study Protocol.
Brief Title: PROFRUVE Program to Promote Fruit and Vegetables Intake Among Children.
Acronym: PROFRUVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Principal Investigator, Victor Manuel Rodriguez Rivera, Doctor, University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: US14/15
Record Dates: First submitted 2017-12-21; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Eating Behavior; Healthy Diet; Fruit and Vegetable Intake; Childhood Obesity
MeSH Terms: conditions — Feeding Behavior; Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group received 14 sessions (one every 15 days) of one hour in the classroom, to work TPB constructs: attitude; subjective norms; perceived behavioural control and intention.
  Interventions: Behavioral: Program based on the theory of planned behaviour
- Control (No Intervention): 2 session of 1 hour each to give general information about fruit and vegetables intake and health.

INTERVENTIONS:
Behavioral: Program based on the theory of planned behaviour — 14 sessions of one hour to work TPB constructs: attitude, subjective norms, perceived behavioural control and intention.
  Arms: Intervention

SUMMARY:
Because fruit and vegetables (FV) intake of children of Vitoria city is low, a controlled intervention program was proposed at school level. The intervention was based on the Theory of Planned Behavior (TPB) as long as behavioral theories have been proved to be the most effective changing infant FV intake pattern. The main purpose of the study is to evaluate the effectiveness of an intervention program based on TPB and aimed to increase FV consumption in schoolchildren aged 8 to 10. For that aim, eligible classrooms from different schools were randomly assigned to the intervention (n=86) or control (n=86) group. The intervention group received 14 sessions of 60 minutes during 9 months of an academic year. Sessions, designed by a multidisciplinary team, are based on TPB and aimed to modify determinants of behavior (attitudes, subjective norms, perceived behavioral control, intention of consumption), and intake of FV itself. Change in fruit and vegetable intake and determinants of eating behavior were evaluated at 9 months of intervention using validated surveys, 7 day food records, 24 hour reminders and questionnaires. This study will provide a valid and useful tool to achieve changes in the consumption of FV at school level. A negative result will be useful to help redefining new strategies in the framework of changing habits in the consumption of FV.

DETAILED DESCRIPTION:
In Vitoria, only two out of ten children and adolescents (aged 6 to 17) consume the recommended three servings of fruit and only one out of ten the recommended two servings of vegetables per day. Average intake of fruit was 1.8 servings/day and 0.8 servings/day for vegetables. For that reason, promotion of the adequate intake of FV must be a priority objective in the promotion of healthy eating habits. One of the most used theories in this type of interventions is TPB (Theory of Planned Behavior). According to this theory, eating behavior and intention of consumption determinants are both personal and environmental. Specifically, the TPB states that attitude, subjective norms and perceived control are determinants that influence both the intention to consume food and the action of consuming it.

The hypothesis of the study is that an intervention program based on theories of behavior and aimed to increase FV intake in schoolchildren aged 8 to 10, will produce changes in attitude, subjective norms, perceived behavioral control and intention of eating fruit and vegetable among children, which in turn will modify the behavior, increasing FV intake.

The main objective of this study is to evaluate the effectiveness of an intervention program based on behavioral theory and aimed to increase FV intake in schoolchildren aged 8 to 10 (short and long effect).

Secondary objectives of the study are (i) to evaluate the change on FV intake on the study population after intervention, (ii) to examine the impact of the intervention program on behavioral determinants, (iii) to analyze the association of the determinants of behavior on FV intake, and (iv) to study the influence between social demographic variables and the effectiveness of the program.

The recruitment of participants begun in may 2015 and they were randomly assigned to intervention or control groups. The intervention group received 14 sessions (one every 15 days) of one hour to work TPB constructs: attitude; subjective norms; perceived behavioural control and intention.

ELIGIBILITY:
Inclusion Criteria:

* all schools with children aged 7-11 years old
* schools with orchard

Exclusion Criteria:

* special schools
* schools carrying out other healthy eating programs at the intervention period

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 230 (Actual)
Dates: Start 2015-05-11 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
FV intake | Change from baseline food and vegetable intake at 9 months of intervention
  Fruit and vegetable daily intake (servings/day)

SECONDARY OUTCOMES:
Eating behaviour determinant: Attitude | Change from baseline attitude at 9 months of intervention
  Evolution of attitude related to eat more FV (1-5 point score, from totally disagree to totally agree)
Eating behaviour determinant: Subjective Norms | Change from baseline subjective norms at 9 months of intervention
  Evolution of subjective norms or social pressure related to eat more FV (1-5 point score, from totally disagree to totally agree)
Eating behaviour determinant: Perceived Behavioural Control | Change from baseline perceived behavioural control at 9 months of intervention
  Evolution of perceived behavioural control related to eat more FV (1-5 point score, from totally disagree to totally agree)
Eating behaviour determinant: Intention | Change from baseline intention at 9 months of intervention
  Evolution of intention of eating more FV (1-5 point score, from totally disagree to totally agree)
Social demographic outcomes | Change from baseline social demographic outcomes at 9 months of intervention
  Participants families social and demographic data
Parents FV intake | Change from parent's baseline food and vegetable intake at 9 months of interventions
  Parents fruits and vegetables daily intake (servings/day)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

REFERENCES:
- [Derived] Arrizabalaga-Lopez M, Rada-Fernandez de Jauregui D, Portillo MDP, Mauleon JR, Martinez O, Etaio I, Tormo-Santamaria M, Bernabeu-Maestre J, Rodriguez VM. A theory-based randomized controlled trial in promoting fruit and vegetable intake among schoolchildren: PROFRUVE study. Eur J Nutr. 2020 Dec;59(8):3517-3526. doi: 10.1007/s00394-020-02185-5. Epub 2020 Feb 1. PMID 32008063
- [Derived] Arrizabalaga-Lopez M, Rada-Fernandez de Jauregui D, Portillo MP, Martinez O, Etaio I, Mauleon JR, Echevarria E, Gomez F, Rodriguez VM. A randomised controlled trial of a program based on the theory of planned behavior to promote fruit and vegetable intake among schoolchildren: PROFRUVE study protocol. BMC Public Health. 2018 Jul 4;18(1):827. doi: 10.1186/s12889-018-5748-3. PMID 29973190